CLINICAL TRIAL: NCT02706821
Title: An Eight-week, Randomized, Double-blind, Placebo-controlled Crossover Clinical Trial of Persimmon Leaf Extract on Anti-diabetes
Brief Title: Anti-diabetic Effects of Persimmon Leaf Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Professor, Chonbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: WJG-HG-PLE
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Prediabetes
Keywords: prediabetes; blood glucose; clinical trial
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment sequence 1 (Active Comparator): PLE (persimmon leaf extract) once a day during 8 weeks cross-over to placebo once a day during 8 weeks.
  Interventions: Dietary Supplement: Persimmon leaf extract; Dietary Supplement: Placebo
- Treatment sequence 2 (Active Comparator): Placebo once a day during 8 weeks cross-over to PLE once a day during 8 weeks.
  Interventions: Dietary Supplement: Persimmon leaf extract; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Persimmon leaf extract — Persimmon leaf extract (PLE), crossover design
Dietary Supplement: Placebo — Placebo, crossover design

SUMMARY:
The investigators performed a 8-week, randomized, double-blind, placebo-controlled crossover human trial to evaluate the efficacy and safety of persimmon leaf extract on blood glucose. The investigators measures changes in diabetes associated parameters, including fasting blood glucose, postprandial blood glucose, insulin, C-peptide and HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years
* Fasting blood glucose (FPG) 100~140 mg/dL or postprandial blood glucose (PPG) 140~250 mg/dL

Exclusion Criteria:

* FPG more than 140 mg/dL
* 2h PPG more than 200 mg/dL
* Type 1 diabetes or HbA1c more than 9.0%
* treatment with corticosteroids within the past 4 weeks
* cardiovascular disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial plasma glucose | baseline day 57, 85 and 141

SECONDARY OUTCOMES:
Fasting plasma insulin | baseline and day 57, 85 and 141
C-peptide | baseline and day 57, 85 and 141
Glycated hemoglobin (HbA1c) | baseline and day 57, 85 and 141
adiponectin | baseline and day 57, 85 and 141
leptin | baseline and day 57, 85 and 141
resistin | baseline and day 57, 85 and 141
Markers of Inflammation | baseline and day 57, 85 and 141
Tumor necrosis factor alpha (TNF-α) | baseline and day 57, 85 and 141
Interleukin-6 (IL-6) | baseline and day 57, 85 and 141
Monocyte chemoattractant protein-1 (MCP-1) | baseline and day 57, 85 and 141